CLINICAL TRIAL: NCT01268709
Title: Effect of Doxepin and Nortriptyline on Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Qom University of Medical Sciences (Other)
Collaborators: Young Researchers Club (Unknown)
Purpose: Treatment
Other Study IDs: YRC-1246
Record Dates: First submitted 2010-12-30; First posted 2010-12-31 (Estimated); Last update posted 2010-12-31 (Estimated); Status verified 2010-12

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Doxepin; Nortriptyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- doxepin (Active Comparator)
  Interventions: Drug: Doxepin
- nortriptyline (Active Comparator)
  Interventions: Drug: Nortriptyline
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Doxepin
  Arms: doxepin
Drug: Nortriptyline
  Arms: nortriptyline
Drug: placebo
  Arms: placebo

SUMMARY:
The objective of this randomized triple blind controlled trial is to compare the effects of Doxepin and Nortriptyline on diarrhea predominant irritable bowel syndrome. In this stuy, 75 patients with IBS are randomly assigned to receive Doxepin , Nortriptyline or placebo, a tablet per day, orally, for two months. Abdominal pain, mucus in the stool, incomplete evacuation, and bloating are measured and compared between groups at the baseline and one and two month after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Presence of diarrhea predominant irritable bowel syndrome according to ROME criteria

Exclusion Criteria:

* Gastrointestinal bleeding
* More than 5% weight loss in the last 6 months
* Presence of any finding in favor of organic disorders in the lab tests or organic disorder in colonoscopy of high risk patients

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Gastrointestinal Research center,Beheshti Hospital, Qom, Qom Province, Iran